CLINICAL TRIAL: NCT05496283
Title: The Effect of Using Denture Adhesives on Patient Satisfaction With Complete Dentures; A Randomized Clinical Trial
Brief Title: Effect of Denture Adhesives on Complete Denture Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Dr. Nadia Ereifej, Associate Professor, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NSEreifej
Record Dates: First submitted 2022-08-07; First posted 2022-08-11 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Complete Edentulism
Keywords: Complete dentures; Patient satisfaction; denture adhesives
MeSH Terms: conditions — Patient Satisfaction | interventions — Dental Cements

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Corega (Experimental): Complete denture patients given Corega denture adhesive.
  Interventions: Other: denture adhesive
- OlivaFix (Experimental): Complete denture patients given OlivaFix denture adhesive.
  Interventions: Other: denture adhesive
- Sea.Bond (Experimental): Complete denture patients given Sea.Bond denture adhesive.
  Interventions: Other: denture adhesive

INTERVENTIONS:
Other: denture adhesive — After 1 month of using the complete denture with no denture adhesives, patients fill up satisfaction and quality of life forms and given 1 of 3 types of denture adhesive to use for month to compare satisfaction and quality of life forms

SUMMARY:
The effect of using denture adhesives on patient satisfaction with complete dentures; A randomized clinical trial.

The study evaluates the effect of using 3 types of denture adhesives on patient satisfaction and quality of life of complete denture patients

DETAILED DESCRIPTION:
Aims: The aims of this study is to compare patient satisfaction and oral health quality of life without using denture adhesive and using 3 types of denture adhesives.

Materials and Methods: 60 completely edentulous patients attending the University of Jordan hospital seeking new sets of complete dentures will be randomly divided into 3 groups (n=20). At delivery of complete dentures, all patients will be given the dentures with no denture adhesive and will be given review appointments after one month of using the dentures. At review appointment, patients will be asked to rate their overall satisfaction and their satisfaction regarding comfort, retention, stability, and efficiency of mastication and speech on a 100-mm visual analog scale (VAS). Participants also will fill out the oral health impact profile for edentulous patients (OHIP-EDENT) questionnaire. Each group will then be given one type of denture adhesive to use; paste-based Corega denture adhesive (CO), Sea Bond maxillary and mandibular denture adhesive strips (SB) and oil-based Olivafix denture adhesive (OF). Patients will be given instructions on how to use each type of adhesive and will be provided with sufficient amount for 1 month. After 1 month, patients will be asked to fill out the same forms

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking new conventional complete dentures for first time
* Patients aged 40-85 years
* Must be completely edentulous for at least 6 months
* Must have well-developed to moderately resorbed maxillary and mandibular ridges
* Must have no denture fissuratum or any traumas from previous dentures
* Must be able to complete and sign the consent form

Exclusion Criteria:

* Patients with relevant medical issues, disorders of masticatory system, neuromuscular dysfunction, auditory problems, psychological or psychiatric conditions that can affect response to treatment
* Patients with oral pathology, xerostomia, or tied tongue condition.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction form | 1 month after denture delivery
  10 aspects regarding patient satisfaction with dentures on 100mm visual analogue scale, with 0 value being completely unsatisfied and 100 for completely satisfied
oral health impact profile for edentulous patients (OHIP-EDENT) | I month after denture delivery
  20 aspects linking the dentures with patient quality of life, with a range of values from 1 to five for each aspect, with 1 being the best and 5 being the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Ereifej, PhD, Principal Investigator — The University of Jordan
Locations (1):
- The University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ereifej NS, Oweis YG, Abu-Awwad M. The effect of using denture adhesives on patient satisfaction with complete dentures; a randomized clinical trial. BMC Oral Health. 2023 Dec 19;23(1):1027. doi: 10.1186/s12903-023-03757-7. PMID 38114958